CLINICAL TRIAL: NCT05986942
Title: Evaluation of the Postoperative Agitation Prevention and Analgesic Efficacy of Perioperative Dexmedetomidine Infusion in a Pediatric Patient Group to Undergo Tonsillectomy and Adenoidectomy
Status: Completed | Type: Observational
Sponsor: Burak Omur (Other)
Responsible Party: Sponsor-Investigator, Burak Omur, assistant professor, Medipol University
Organization: Medipol University (Other)
Other Study IDs: 000030195314317
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Anxiety; Postoperative Pain; Bleeding
Keywords: Dexmedetomidine; tonsillectomy; adenoidectomy; postoperative anxiety
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative; Hemorrhage | interventions — Fentanyl; Dexmedetomidine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dex: patients using dexmedetomidine infusion
  Interventions: Drug: Dexmedetomidine
- Fen: patients using fentanyl for induction
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — In Group dex, dexmedetomidine infusion will be administered to the patient during the operation. Fentanyl bolus dose will be administered during anesthesia induction in group Fen.
  Other Names: Talinat
  Groups: Fen
Drug: Dexmedetomidine — In Group dex, dexmedetomidine infusion will be administered to the patient during the operation. Fentanyl bolus dose will be administered during anesthesia induction in group Fen.
  Other Names: Precedex
  Groups: Dex

SUMMARY:
Dexmedetomidine is a drug known for its pain-relieving and restlessness-reducing effects. The purpose of this run is to use the association between this use during surgery and the attrition of post-operative pain and discomfort. In the research, laboratory and monitoring results will be obtained before, during and after the operation. Postoperative patient complaints will be evaluated at the postoperative service visit. This study is decided on a completely voluntary basis.

ELIGIBILITY:
Inclusion Criteria:

Patients with ASA 1-2, aged 2-10 years, scheduled for elective tonsillectomy and/or adenoidectomy operation will be included.

Exclusion Criteria:

developmental delay anxiety disorder Known history of allergy to alpha-2 agonistic agents use of antipsychotic medication beta blocker use of anticonvulsant drugs chronic pain syndrome with cardiac and craniofacial anomalies

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with ASA 1-2, aged 2-10 years, scheduled for elective tonsillectomy and/or adenoidectomy operation will be included
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
postoperative pain | Pain was evaluated at 0, 2, 4, 6 and 8 hours postoperatively.
  Postoperative pain level will be measured using the FLACC pain scale (face, legs, activity, cry, consolability). 4 and above will be considered as high pain level, below 4 as low pain level.
postoperative anxiety | anxiety was evaluated at 0, 2, 4, 6 and 8 hours postoperatively.
  Postoperative anxiety level will be measured using the Pediatric Anesthesia Emergence Delirium Scale (PAED). A value of 12 and above will be considered high anxiety, and values below 12 will be considered low anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Yaşar G Gül, Study Director — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Patel A, Davidson M, Tran MC, Quraishi H, Schoenberg C, Sant M, Lin A, Sun X. Dexmedetomidine infusion for analgesia and prevention of emergence agitation in children with obstructive sleep apnea syndrome undergoing tonsillectomy and adenoidectomy. Anesth Analg. 2010 Oct;111(4):1004-10. doi: 10.1213/ANE.0b013e3181ee82fa. Epub 2010 Aug 12. PMID 20705788
- [Result] Lin R, Ansermino JM. Dexmedetomidine in paediatric anaesthesia. BJA Educ. 2020 Oct;20(10):348-353. doi: 10.1016/j.bjae.2020.05.004. Epub 2020 Jul 22. No abstract available. PMID 33456916